CLINICAL TRIAL: NCT01058746
Title: A Prospective Randomized Controlled Clinical Trial of Restrictive Versus Liberal Perioperative Fluid Management for Patients Undergoing Pancreatic Resection
Brief Title: Randomized Trial of Restrictive Versus Liberal Perioperative Fluid Management for Patients Undergoing Pancreatic Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-185
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; surgery; Pancreaticoduodenectomy; Central Pancreatectomy; Distal Pancreatectomy; resection; IV fluids; 09-185
MeSH Terms: conditions — Pancreatic Neoplasms

ARMS (2):
- pts undergoing pancreatic resection Restrictive arm (Active Comparator): All patients will receive Normosol or equivalent solution, 0.5 ml/kg/fasted hour IV (approximately from 8am to time of induction) during induction of anesthesia. All patients will then receive maintenance fluids consisting of Normosol or equivalent solution at 6 ml/kg/operative hour. After randomization occurs, those patients randomized to the Restricted Arm will continue to receive Normosol or equivalent solution at 6ml/kg/operative hour.
  Interventions: Other: restrictive perioperative fluid management
- pts undergoing pancreatic resection Liberal arm (Active Comparator): All patients will receive Normosol or equivalent solution, 0.5 ml/kg/fasted hour IV (approximately from midnight to time of induction) during induction of anesthesia. All patients will then receive maintenance fluids consisting of Normosol or equivalent solution at 6 ml/kg/operative hour. Those patients randomized to the Liberal Arm will receive an additional Normosol bolus or equivalent solution equal to (another) 1.5 ml/kg/fasted hour IV (to bring the total to 2 ml/kg/fasted hour) plus an additional bolus of Normosol or equivalent solution 6ml/kg/operative hour to bring the hourly rate to 12ml/kg/operative hour with a maximum of 1000 ml/operative hour.
  Interventions: Other: Liberal perioperative fluid management

INTERVENTIONS:
Other: restrictive perioperative fluid management — Normosol or equivalent solution 0.5 ml/kg/fasted hour IV (8am to time of induction) during induction of Anesthesia. Maintenance IV Normosol or equivalent solution at 6 ml/kg/operative hour. Blood loss to be replaced volume: volume with colloid until transfusion criteria met. Additional fluid boluses of 100ml Normosol or equivalent solution or bolus pressors (phenylephrine 40mcg or ephedrine 5mg) at the discretion of the Anesthesiologist to maintain patient hemodynamic stability.
  Arms: pts undergoing pancreatic resection Restrictive arm
Other: Liberal perioperative fluid management — Normosol or equivalent solution 0.5 ml/kg/fasted hr IV (8am to time of induction) of Anesthesia. Maintenance IV Normosol or equiv solution at 6 ml/kg/oper hr. At randomiz to the Liberal arm in the OR, an addit bolus of Normosol or equiv solution 1.5 ml/kg/fasted hr IV (8am to time of induction) will be given to bring the total to Normosol or equiv solution 2ml/kg/fasted hr IV (8am to time of induction). Pt will get an addit bolus of Normosol or equivalent solution 6ml/kg/oper hr. Maintenance IV Normosol or equivalent solution will then commence at 12ml/kg/operative hr with maximum of 1000 ml/operative hr. Blood loss replaced volume: with colloid, until transfusion criteria met (Additional fluid boluses of 100ml Normosol or equivalent solution or bolus pressors (phenylephrine 40mcg or ephedrine 5mg) used at the discretion of the Anes to maintain pt hemodynamic stability. Addit fluid boluses of 250ml Normosol or equivalent solution for urine output less than 1ml/kg for 2 hrs.
  Arms: pts undergoing pancreatic resection Liberal arm

SUMMARY:
The purpose of this study is to help us learn what the best amount of fluid is that patients should receive during pancreas surgery. Patients will receive either the liberal fluid amount for this surgery or a restricted fluid amount.

Both amounts of fluid have been used safely in patients having similar surgeries. These amounts have not been compared in pancreatic surgery. The fluids regimens that will be given are not experimental.

This study will compare patients in the liberal and restricted fluid groups in terms of the nature of any surgical complications (problems)and recovery from surgery, including length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Adults > or = 18 years
* Patients scheduled for Pancreaticoduodenectomy, Central Pancreatectomy or Distal Pancreatectomy.

Exclusion Criteria:

* Pregnancy
* History of active coronary disease unless a cardiac stress test showing no reversible ischemia and normal LV function within 30 days of operation
* MI within 3 months
* History of stroke
* History of congestive heart failure and ejection fraction less than 35%
* History of severe COPD and resting oxygen saturation (SpO2) < 90%
* Renal dysfunction (Cr > 1.8)
* Abnormal coagulation parameters (INR > 1.5 not on Coumadin, or platelet
* Presence of active infection including HIV
* BMI > 35
* American Society of Anesthesiologists Status > III, assigned at time of preoperative visit
* Corticosteroid use > 10 mg Prednisone/day
* Bilirubin > 10.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
To determine if restrictive perioperative fluid management results in fewer complications, morbidity and decreased length of stay in patients undergoing pancreatic resection, compared to liberal fluid management. | 3 years

SECONDARY OUTCOMES:
Determine if restrictive perioperative fluid management, comp to liberal periop fluid management, decreases delayed gastric emptying, length of stay (LOS) & the incidence of other, less frequent morbidity in adult patients getting pancreatic resection. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Florence Grant, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm